CLINICAL TRIAL: NCT01966003
Title: A Randomized, Double-blind, Phase 3 Study Evaluating the Efficacy and Safety of ABP 215 Compared With Bevacizumab in Subjects With Advanced Non-Small Cell Lung Cancer
Brief Title: Efficacy and Safety Study of ABP 215 Compared With Bevacizumab in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120265; 2013-000738-36 (EudraCT Number)
Record Dates: First submitted 2013-10-04; First posted 2013-10-21 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Non-small Cell Lung Cancer Metastatic
MeSH Terms: interventions — Carboplatin; Paclitaxel; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABP 215 (Experimental): Participants received 15 mg/kg ABP 215 administered as an intravenous (IV) infusion every 3 weeks (Q3W) for 6 cycles and carboplatin and paclitaxel chemotherapy Q3W for at least 4 and not more than 6 cycles.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: ABP 215
- Bevacizumab (Active Comparator): Participants received bevacizumab 15 mg/kg administered as an intravenous (IV) infusion every 3 weeks (Q3W) for 6 cycles and carboplatin and paclitaxel chemotherapy Q3W for at least 4 and not more than 6 cycles.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Carboplatin — Administered at an area under the concentration-time curve (AUC) 6 by IV infusion Q3W
  Other Names: Paraplatin
Drug: Paclitaxel — Administered 200 mg/m² IV Q3W
  Other Names: Taxol
Drug: ABP 215 — Administered 15 mg/kg Q3W by IV infusion
  Arms: ABP 215
Drug: Bevacizumab — Administered 15 mg/kg Q3W by IV infusion
  Other Names: Avastin
  Arms: Bevacizumab

SUMMARY:
The purpose of this research study is to compare the effectiveness and safety of ABP 215 against bevacizumab in men and women with advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-squamous non-small cell lung cancer (NSCLC)
* Subjects must be initiating first-line carboplatin/paclitaxel chemotherapy within 8 days after randomization and expected to receive at least 4 cycles of chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1

Exclusion Criteria:

* Small cell lung cancer (SCLC) or mixed SCLC and NSCLC
* Central nervous system (CNS) metastases
* Malignancy other than NSCLC
* Palliative radiotherapy for bone lesions inside the thorax
* Prior radiotherapy of bone marrow
* Known to be positive for hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
* Life expectancy < 6 months
* Woman of child-bearing potential who is pregnant or is breast feeding or who is not consenting to use highly effective methods of birth control during treatment and for an additional 6 months after the last administration of the protocol specified treatment
* Man with a partner of childbearing potential who does not consent to use highly effective methods of birth control during treatment and for an additional 6 months after the last administration of the protocol specified treatment
* Subject has known sensitivity to any of the products to be administered during the study, including mammalian cell derived drug products
* Other inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2015-07-23 (Actual); Study Completion 2015-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- Research Site, Bismarck, North Dakota, United States
- Research Site, Fremantle, Western Australia, Australia
- Bulgaria (2):
  - Research Site, Veliko Tarnovo, Veliko Tarnovo
  - Research Site, Rousse

REFERENCES:
- [Derived] Thatcher N, Goldschmidt JH, Thomas M, Schenker M, Pan Z, Paz-Ares Rodriguez L, Breder V, Ostoros G, Hanes V. Efficacy and Safety of the Biosimilar ABP 215 Compared with Bevacizumab in Patients with Advanced Nonsquamous Non-small Cell Lung Cancer (MAPLE): A Randomized, Double-blind, Phase III Study. Clin Cancer Res. 2019 Apr 1;25(7):2088-2095. doi: 10.1158/1078-0432.CCR-18-2702. Epub 2019 Jan 7. PMID 30617139
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 101 sites (14 sites in the US, 11 in Russia, 10 in Australia, 9 in Germany, 8 in Poland, 7 in Hungary, 7 in Romania, 6 in Italy, 6 in Spain, 5 in Bulgaria, 5 in Greece, 3 in the Czech Republic, 3 in Mexico, 3 in Taiwan, 2 in the Netherlands, 1 in Canada, and 1 in Hong Kong).
Pre-assignment Details: Eligible participants were randomized in a 1:1 ratio to receive ABP 215 or bevacizumab. Participants were stratified by geographic region (Eastern Europe vs Western Europe vs Asia Pacific/Other vs North America), Eastern Cooperative Oncology Group (ECOG) performance status (0 vs 1), and sex.
Period: Overall Study
Arm/Group | ABP 215 | Bevacizumab
Started | 328 | 314
Received Study Drug | 324 | 309
Completed | 58 | 44
Not Completed | 270 | 270
Not completed — Death | 43 | 36
Not completed — Protocol Violation | 6 | 4
Not completed — Lost to Follow-up | 4 | 3
Not completed — Physician Decision | 12 | 13
Not completed — Withdrawal by Subject | 29 | 19
Not completed — Plan to Receive Other Anticancer Therapy | 131 | 127
Not completed — Plan to Receive Commercial Bevacizumab | 44 | 67
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABP 215 | Bevacizumab | Total
Number analyzed (Participants) | 328 | 314 | 642
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.09) | 61.6 (8.88) | 61.6 (8.98)
Age, Customized [Number; unit: participants]
  < 65 years | 199 | 191 | 390
  ≥ 65 years | 129 | 123 | 252
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 126 | 258
  Male | 196 | 188 | 384
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 16 | 30
  Not Hispanic or Latino | 314 | 298 | 612
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Participants were allowed to choose multiple races.
  participants
    White | 315 | 300 | 615
    Black or African American | 2 | 5 | 7
    Asian | 6 | 7 | 13
    American Indian or Alaska Native | 2 | 0 | 2
    Native Hawaiian or other Pacific Islander | 1 | 0 | 1
    Other | 4 | 2 | 6
Geographic Region [Number; unit: participants]
  Eastern Europe | 189 | 186 | 375
  Western Europe | 78 | 76 | 154
  North America | 31 | 26 | 57
  Asia Pacific/Other | 30 | 26 | 56
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  participants
    Grade 0 | 127 | 117 | 244
    Grade 1 | 201 | 197 | 398

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Objective Response
Description: Tumor assessments were performed by central, independent, blinded radiologists according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 using computed tomography (CT) or magnetic resonance imaging (MRI) scans of the chest and abdomen. Objective response is defined as a best overall response of partial response (PR) or complete response (CR) as defined by RECIST v1.1. All participants who did not meet the criteria for CR or PR by the end of the study were considered non-responders.
  CR: Disappearance of all target and non-target lesions and no new lesions. Any pathological lymph nodes must be reduced in short axis to < 10 mm.
  PR: Disappearance of all target lesions with persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits, and no new lesions, or, at least a 30% decrease in the sum of diameters of target lesions, with no progression of existing non-target lesions and no new lesions.
Time Frame: Disease assessments were performed at weeks 1, 7, 13, 19, and approximately every 9 weeks thereafter. The mean actual follow-up time from randomization was 4.7 and 5.0 months for ABP 215 and bevacizumab, respectively.
Population: Intent-to-treat population which consisted of all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | ABP 215 | Bevacizumab
Number analyzed (Participants) | 328 | 314
percentage of participants | 39.0 | 41.7
Statistical Analysis 1: Comparison: ABP 215 vs Bevacizumab; The risk ratio (ABP 215/Bevacizumab) and 90% confidence interval (CI) were estimated using a generalized linear model adjusted for the stratification factors (region, sex, and ECOG performance status); Test type: Non-Inferiority or Equivalence — Clinical equivalence of the primary endpoint was demonstrated by comparing the 2-sided 90% CI of the risk ratio in objective response rate between ABP 215 and bevacizumab with an equivalence margin of (0.67, 1.5); Risk Ratio (RR) = 0.93, 90% CI 2-sided [0.80 to 1.09]
Statistical Analysis 2: Comparison: ABP 215 vs Bevacizumab; Risk difference (ABP 215 - Bevacizumab) and 90% CI were estimated using a generalized linear model adjusted for the randomization stratification factors geographic region, ECOG performance status, and sex; Test type: Superiority or Other; Risk Difference (RD) = -2.90, 90% CI 2-sided [-9.26 to 3.45]

2. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was calculated as the time from the first objective response (PR or CR) to disease progression per RECIST v1.1 based on the central, independent, blinded radiologists' review.
  DOR was only calculated for participants with an objective response. For responders not meeting the criterion for progression by the end of the study, DOR was censored at the date of the last evaluable tumor assessment.
  Progressive Disease was defined as at least a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 mm, or, unequivocal progression of existing non-target lesions, or any new lesions.
Time Frame: as for outcome 1
Population: Intent-to-treat population with an objective response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABP 215 | Bevacizumab
Number analyzed (Participants) | 128 | 131
months | 5.8 [4.9 to 7.7] | 5.6 [5.1 to 6.3]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from the randomization date to the date of disease progression using RECIST v1.1 based on the central, independent, blinded radiologists' review, or death. Participants who were alive and did not meet the criteria for progression by the end of the study were censored at their last evaluable disease assessment date. Participants with no evaluable tumor assessments after randomization who did not die by the end of the study were censored on the randomization date.
  Progressive Disease was defined as at least a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 mm, or, unequivocal progression of existing non-target lesions, or any new lesions.
Time Frame: From randomization until the end of study; The mean actual follow-up time from randomization was 4.7 and 5.0 months for ABP 215 and bevacizumab, respectively.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABP 215 | Bevacizumab
Number analyzed (Participants) | 328 | 314
months | 6.6 [6.3 to 7.9] | 7.9 [6.6 to 8.2]
Statistical Analysis 1: Comparison: ABP 215 vs Bevacizumab; The hazard ratio for ABP 215 relative to bevacizumab was based on a stratified Cox proportional hazards model. Stratification factors are geographic region, ECOG performance status, and sex; Test type: Superiority or Other; Hazard Ratio (HR) = 1.03, 90% CI 2-sided [0.83 to 1.29]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4, and according to the following scale: Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Death due to AE.
  A serious adverse event (SAE) is defined as an AE that meets at least 1 of the following serious criteria:
  * fatal
  * life-threatening
  * required inpatient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event
Time Frame: up to 19 weeks
Population: Safety analysis population consisted of all participants who received any amount of study drug.
Measure: Number; unit: participants
Arm/Group | ABP 215 | Bevacizumab
Number analyzed (Participants) | 324 | 309
participants
  Any adverse event | 308 | 289
  Any grade ≥ 3 adverse event | 139 | 137
  Any fatal adverse event | 13 | 11
  Any serious adverse event | 85 | 71
  Any AE leading to discontinuation of study drug | 61 | 53
  Any AE leading to discontinuation of chemotherapy | 74 | 59
  Any AE leading to dose delay of study drug | 73 | 69
  Any AE leading to dose delay of any chemotherapy | 86 | 83
  Any AE leading to dose reduction of chemotherapy | 48 | 49

5. Secondary Outcome: Number of Participants Who Developed Anti-drug Antibodies
Description: Two validated assays were used to detect the presence of anti-ABP 215 antibodies. Samples were first tested in an electrochemiluminescence (ECL)- based bridging immunoassay to detect antibodies capable of binding to ABP 215 (Binding Antibody Assay). Samples confirmed to be positive for binding antibodies were subsequently tested in a non-cell based target binding assay to determine neutralizing activity against ABP 215 (Neutralizing Antibody Assay). If a post-dose sample was positive for binding antibodies and demonstrated neutralizing activity at the same time point, the sample was defined as positive for neutralizing antibodies.
Time Frame: 44 weeks (6 months after end of treatment)
Population: Safety analysis population with available data
Measure: Number; unit: participants
Arm/Group | ABP 215 | Bevacizumab
Number analyzed (Participants) | 294 | 284
participants
  Binding antibody positive | 4 | 7
  Neutralizing antibody positive | 0 | 0

6. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from the randomization date to date of death. Participants alive at the end of study were censored at the last date known to be alive, derived from dates collected within the study that implied a participant was alive.
  Participants were followed for survival status during the treatment phase and thereafter every 9 weeks until the end of the clinical study, consent was withdrawn, they were lost to follow-up, died, or had proscribed therapy (eg, commercial bevacizumab, non-study anti-cancer treatment).
Time Frame: as for outcome 3
Population: Safety analysis population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABP 215 | Bevacizumab
Number analyzed (Participants) | 324 | 309
months | NA [NA to NA] — Could not be estimated due to the low number of deaths | NA [14.6 to NA] — Could not be estimated due to the low number of deaths
Statistical Analysis 1: Comparison: ABP 215 vs Bevacizumab; Hazard ratio for ABP 215 relative to bevacizumab, based on a stratified Cox proportional hazards model. Stratification factors are geographic region, ECOG performance status, and sex; Test type: Superiority or Other; Hazard Ratio (HR) = 1.10, 90% CI 2-sided [0.75 to 1.61]

ADVERSE EVENTS:
Time Frame: 19 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | ABP 215 | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 85/324 | 71/309
Other Adverse Events (participants affected / at risk) | 286/324 | 276/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABP 215 (N=324) | Bevacizumab (N=309)
Anaemia (Blood and lymphatic system disorders) | 3 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 8
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 6 | 3
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Paroxysmal arrhythmia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Mesenteric artery embolism (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Death (General disorders) | 2 | 1
Fatigue (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 2 | 2
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Sudden death (General disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Abscess soft tissue (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cytomegalovirus hepatitis (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 2
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Neutropenic infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 2
Pilonidal cyst (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 5
Pseudomonas infection (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 2 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 1
Hallucinations, mixed (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Prophylaxis (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Embolism arterial (Vascular disorders) | 1 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABP 215 (N=324) | Bevacizumab (N=309)
Anaemia (Blood and lymphatic system disorders) | 65 | 60
Leukopenia (Blood and lymphatic system disorders) | 23 | 23
Neutropenia (Blood and lymphatic system disorders) | 55 | 60
Thrombocytopenia (Blood and lymphatic system disorders) | 47 | 43
Constipation (Gastrointestinal disorders) | 36 | 36
Diarrhoea (Gastrointestinal disorders) | 39 | 55
Gingival bleeding (Gastrointestinal disorders) | 9 | 19
Nausea (Gastrointestinal disorders) | 82 | 95
Stomatitis (Gastrointestinal disorders) | 15 | 18
Vomiting (Gastrointestinal disorders) | 37 | 41
Asthenia (General disorders) | 49 | 42
Fatigue (General disorders) | 57 | 59
Pyrexia (General disorders) | 19 | 20
Weight decreased (Investigations) | 18 | 16
Decreased appetite (Metabolism and nutrition disorders) | 54 | 42
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 19
Bone pain (Musculoskeletal and connective tissue disorders) | 20 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 39 | 44
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 20
Dizziness (Nervous system disorders) | 13 | 25
Headache (Nervous system disorders) | 28 | 24
Neuropathy peripheral (Nervous system disorders) | 56 | 38
Paraesthesia (Nervous system disorders) | 28 | 40
Peripheral sensory neuropathy (Nervous system disorders) | 18 | 16
Polyneuropathy (Nervous system disorders) | 20 | 22
Proteinuria (Renal and urinary disorders) | 26 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 24
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 44 | 39
Alopecia (Skin and subcutaneous tissue disorders) | 140 | 127
Hypertension (Vascular disorders) | 51 | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.